CLINICAL TRIAL: NCT05653154
Title: Preoperative Concerns in Older Adults
Brief Title: Preoperative Survey
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Anesthesiologist, University Health Network, Toronto
Other Study IDs: CAPCR # 22-5163
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment
Keywords: Elderly, surgical
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will examine preoperative concerns in older adults through the use of a self-administered questionnaire. The development of this questionnaire will involve adapting survey questions from previously validated studies, creating new questions, and generating a comprehensive questionnaire.

DETAILED DESCRIPTION:
The primary objective is to assess the preoperative concerns in older adults. This objective will be assessed by using a self-administered questionnaire.

The secondary objective is to examine older adults' attitudes toward preoperative cognitive assessments, functional assessments, and prehabilitation programs. Similarly, this objective will be assessed by using a self-administered questionnaire.

Survey administration will be completed online and in person. Recruited participants will receive an email that contains an external link to the online version of the survey that will be administered on Research Electronic Data Capture (REDCap), an online platform to complete secure surveys. Once received, participants will be able to anonymously complete the survey and not have to provide any identification information except for general sociodemographic variables. Alternatively, study personnel will administer the questionnaire online/ in person at the preoperative clinic to assess surgical population at Mount Sinai Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Older adults, who are aged 65 or older and
* Medical patients in geriatric clinic or surgical inpatients in pre-operative clinics

Exclusion Criteria:

• Lack English language capability

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
preoperative concerns | 1 day
  current daily functional status

SECONDARY OUTCOMES:
Cognitive assessments | 1 day
  Administration of cognitive status questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - 399 Bathurst St., Toronto Western Hospital, Dept. of Anesthesia, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No